CLINICAL TRIAL: NCT00598455
Title: Tuberous Sclerosis Complex Natural History Study: Renal Manifestations
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Loma Linda University (Other); Massachusetts General Hospital (Other); Boston Children's Hospital (Other); University of Alabama at Birmingham (Other); University of Pennsylvania (Other); Connecticut Children's Medical Center (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Other Study IDs: TS0500008; W81XWH-06-1-0538
Record Dates: First submitted 2007-12-27; First posted 2008-01-22 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Tuberous Sclerosis Complex
Keywords: angiomyolipomata; tuberous sclerosis complex
MeSH Terms: conditions — Tuberous Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Eighty percent of patients with tuberous sclerosis complex (TSC) have renal angiomyolipomata. These lesions grow and can lead to significant morbidity by hemorrhage or renal failure. Understanding the natural history of these lesions and understanding which lesions may be more prone to grow quickly or develop aneurysms that predispose to hemorrhage will greatly assist clinical care of patients with TSC. The objective is to test the hypothesis that serial MR and CT imaging will allow objective, reproducible quantification of angiomyolipoma growth by volumetric analysis, and analysis of lesions characteristics will identify angiomyolipomata with rapid growth potential that would require intervention. The specific aim of this proposal is to collect clinically obtained serial abdominal imaging from the Tuberous Sclerosis Natural History Consortium Centers and analyze the volume and adiposity of the individual angiomyolipomata. The growth rate is hypothesized to have an inverse relationship to adiposity. Yearly renal MR or CT imaging will be performed of patients with TSC. The images will be coded at the site of acquisition, and transferred via VPN to a secure server at Cincinnati Children's Hospital Medical Center. Using innovative imaging processing software (Cincinnati Children's Hospital Image Processing Software (CCHIPS), the image data will be segmented to reveal various tissue components based on signal intensities. Different signal intensities can differentiate normal renal parenchyma, and renal angiomyolipomata. Using the imaging data and the novel software, the volume of an individual angiomyolipoma, as well as the adiposity will be determined. Imaging at enrollment (year 1) will serve as baseline. At years two and three, the lesions will undergo repeat analysis. Angiomyolipoma growth rates and adiposity over three years will be analyzed to test the hypothesis above.

DETAILED DESCRIPTION:
Objectives.

Our objective is to test the hypothesis that serial MR and CT imaging will allow objective, reproducible quantification of angiomyolipoma growth by volumetric analysis, and analysis of lesions characteristics will identify angiomyolipomata with rapid growth potential that would require intervention.

The specific aim of this proposal is to collect clinically obtained serial abdominal imaging from the Tuberous Sclerosis Natural History Consortium Centers and analyze the volume and adiposity of the individual angiomyolipomata. The growth rate is hypothesized to have an inverse relationship to adiposity. The prognostic value of identifying lesions with aggressive growth characteristics is very large, and intervention can be instituted early in order to reduce the renal damage.

Study Population.

1. The target population for this study will be patients with tuberous sclerosis who attend a tuberous sclerosis clinic that is part of the consortium. The data collected will include routine imaging data, age, gender, and if know, the genotype. Approximately 855 patients throughout the United States will be asked to participate in this natural history study and 450 of those are anticipated to consent and have complete data on 3 years of CT and MR Imaging Scans to measure angiomyolipoma growth and adiposity.
2. Patients attending the tuberous sclerosis clinics that are members of the consortium will be asked if they would be involved in the study.
3. Imaging will be obtained as part of the standard of care at the Consortium Centers. Imaging done on pregnant patients will not be excluded. MRI has been used now extensively for pregnant patients.

Protocol Design.

This is a natural history study involving the imaging characteristics of angiomyolipomata found in patients with tuberous sclerosis complex. This study offers the potential benefit that the lesion characteristics and growth rate will be monitored. Patel et al. posit that growth rates of greater than 0.5 cm/year for solid tumors are worrisome for malignancy. Patients harboring lesions that exhibit faster growth rates will be identified so that they can be more carefully monitored. During the course of the study, should we detect concerning features, the Consortium Center TS Clinic Director will be alerted. Imaging modalities that may be used include CT scans. The patient data being collected will be done so for clinical reasons, and every effort will be made to use the least possible radiation exposure. There are several ways to reduce the exposure, and these limiting techniques will be employed for each scan. The scans will be performed both pre and post contrast using an agent such as Optiray® so that vascularity can be assessed. Patients may also be imaged with a 1.5 Tesla magnet in a supine position using a phased array torso coil or body coil, depending on patient size. When compatible, respiratory compensation will be used to diminish respiratory artifact. Overall imaging time for the following sequences will be approximately 45 minutes.

a. Recruitment process: Patients will be recruited from patients seen at the Tuberous Sclerosis Natural History Consortium Centers, including Cincinnati Children's Hospital, Loma Linda University, University of Pennsylvania Medical Center, Connecticut Children's Medical Center, Vanderbilt University, Columbus Children's, Texas Scottish Rite Hospital, Massachusetts General Hospital, Miami Children's Hospital, Minnesota Epilepsy Group, Dartmouth University, Washington Children's Hospital, New York University School of Medicine, University of Texas, Houston, Children's Hospital, Boston, and Children's Hospital, Pittsburgh.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive yearly follow-up at their respective tuberous sclerosis clinic. Such clinics have a director who is knows their patients well.
* Patients known to have an angiomyolipoma between the ages of 7-
* 65 years
* Pregnant women to be included if tested with MR

Exclusion Criteria:

* Patients who are not seen annually and therefore do not have yearly imaging.
* Patients who do not have an angiomyolipoma.
* Patients who are not likely to follow-up as recommended.
* Use of an investigational drug, including rapamycin, within the last 30 days.
* Pregnant women to be excluded if they cannot be tested with MR

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: a. The target population for this study will be patients with tuberous sclerosis who attend a tuberous sclerosis clinic that is part of the consortium. The data collected will include routine imaging data, age, gender, and if know, the genotype. Approximately 855 patients throughout the United States will be asked to participate in this natural history study and 450 of those are anticipated to consent and have complete data on 3 years of CT and MR Imaging Scans to measure angiomyolipoma growth and adiposity.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2008-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Bissler, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's, Cincinnati, Ohio, United States